CLINICAL TRIAL: NCT05091489
Title: Qualitative Assessment About PrEP Acceptability in Key-populations and Conditions Required for Community-based PrEP Implementation in Cambodia
Brief Title: ANRS 12415 - Quali PrEP Cambodia
Acronym: ANRS 12415
Status: Completed | Type: Observational
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: University of Health Sciences, Phnom Penh, Cambodia (Unknown); National Center for HIV/AIDS Dermatology and STDs, Phnom Penh, Cambodia (Unknown)
Responsible Party: Principal Investigator, Marion Fiorentino, Principal Investigator, Institut de Recherche pour le Developpement
Other Study IDs: PREP2021-MF
Record Dates: First submitted 2021-09-23; First posted 2021-10-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hiv
Keywords: Men who have sex with men (MSM); Transgender women (TGW); Sex workers; Healthcare; Community-based organisations; PrEP; Pre-exposition prophylaxis; focus group; interview; Cambodia; qualitative; acceptability; prevention; men who have sex with men; decision makers; community workers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (16):
- Men who have sex with men (MSM) non-using PrEP: Focus group (10 persons)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Male entertainment workers: Focus group (10 persons)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Free-lance based entertainment female workers non-using PrEP: Focus group (10 persons)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Venue-based entertainment female workers non-using PrEP: Focus group (10 persons)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Transgender women (TGW) non-using PrEP: Focus group (10 persons)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Healthcare workers in charge of key-populations: Focus group (10 persons)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Community workers in charge of key-populations: Focus group (10 persons)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- PrEP users: Focus group (10 persons)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- NCHADS: Individual semi-directive interview (1 person) (NCHADS: operational unit of the Ministry of Health in charge of health sector policy development for HIV/AIDS)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- National Aids Authority: Individual semi-directive interview (1 person) (National Aids Authority: in charge to lead, manage, coordinate and facilitate the comprehensive and multi-sectoral response to HIV and AIDS in Cambodia)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Ministry of Health: Individual semi-directive interview (1 person)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Key influencer in the MSM and/or TGW community: Individual semi-directive interview (1 person)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Key influencer in the EW community: Individual semi-directive interview (1 person)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Khana: Individual semi-directive interview (1 person)
  Khana : an umbrella organization belonging to the HIV/AIDS international Alliance
  Interventions: Other: Qualitative assessment about PrEP acceptability
- High class and hidden MSM: Individual semi-directive interview (1 person)
  Interventions: Other: Qualitative assessment about PrEP acceptability
- Discontinued PrEP user: Individual semi-directive interview (1 person)
  Interventions: Other: Qualitative assessment about PrEP acceptability

INTERVENTIONS:
Other: Qualitative assessment about PrEP acceptability — Qualitative research among key-populations, community and healthcare workers, and decision and policy makers, including focus group and semi-directive interviews

SUMMARY:
Hypothesis:

* Hypothesis 1 : Regarding the recentness of preexposure prophylaxis (PrEP) implementation with an uptake of 20% and according to the first consultative meeting, awareness and acceptability of PrEP seems to be low in key-populations of Cambodia
* Hypothesis 2 : Individual, social and structural barriers and facilitating factors of PrEP implementation as perceived by health workers and community-based organizations would be similar to what was observed worldwide 4,8.
* Hypothesis 3: Some subgroups of key-populations are difficult to reach in health facilities. Community organizations can play a critical role to provide PrEP information, initiation and counselling with the support of new technologies.
* Hypothesis 4: Community organizations might lack financial, logistical and skill capacities to deliver PrEP in good conditions

Main objective:

• To qualitatively evaluate the knowledge, awareness, perception, experience and acceptability of PrEP among key populations (entertainment workers (EW), men who have sex with men (MSM), transgender women (TW)), and among healthcare and community workers in charge of key populations

Secondary objectives:

* To better understand the characteristics, needs and expectations of community-based organizations (CBOs), in order to define the optimal conditions for community-based PrEP implementation
* To identify tools that could be useful to increase PrEP awareness and acceptability, especially new technologies (apps, websites)

Methodology: Qualitative study Focus groups with key-populations, healthcare and community workers Semi-directive interviews with decision makers and policy makers Estimated enrolment: 10 participants per focus group, 8 focus groups, 80 participants in focus groups, 6 interviewed persons, 86 participants in total

Study population: Men who have sex with men (MSM), entertainment workers (EW), transgender women (TGW), healthcare workers, community workers, decision and policy makers

ELIGIBILITY:
Eligibility criteria for key-populations included in focus groups

* All key-populations

  * Having consented to participate into the research
  * Self-declared negative HIV status
* Men who have sex with men (MSM): being sexually active and having had anal sex with at least one male (including TGW women) partner in the past 12 months.
* Transgender women (TGW): Being biologically male at birth and self-identified as a woman or third gender, reporting having anal sex with at least one male in the past 12 months
* Male entertainment workers (MEW): having at least one sexual intercourse in exchange of money in the last month. MEW are engaged in transactional sex by Facebook, via online App (Grinder, Blue) and massage parlor.
* Female entertainment workers: Venue-based (work in entertainment establishment) or non-venue based (freelance/street-based or park-based) women having at least one sexual intercourse in exchange of money in the last month. Venue-based EW (VEW) are defined as EW engaged in transactional sex for supplementary income which are employees in entertainment venues such as karaokes, bars, beer gardens, massage parlours. Free-lance EW (FEW) are defined as EW engaged in transactional sex in short-time hotel or public parks21 or "high-class" EW working in salons or using apps such as Line. We hypothesized that FEW and VEW have different sex behaviours as well as different perceptions and motivations towards PrEP.
* PrEP users: MSM or TGW who have started medical PrEP in the pilot program "Khmer PrEP" and MSM or TGW who have independently started medical PrEP in private. If possible, individuals who are currently receiving PrEP and individuals who discontinued will be included.

Exclusion criteria for key-populations : self-declared HIV-positive

Eligibility criteria for community and health workers

* Health workers and counselors: 1/ currently working in a HIV service targeting key populations (Samdach Ov Referral Hospital, Meanchey Referral Hospital, Social Health Clinic). 2/ currently working in a health service delivering PrEP (Chhouk Sar Clinic, Pochentong and Chaktomuk hospitals, RHAC)
* Community workers: currently working in CBOs with EW, TG and/or MSM (Cambodian Women for Peace and Development (CWPD), Men's Health Cambodia (MHC), Men's Health Social Service (MHSS)

Individual semi-directive interviews will be conducted:

* NCHADS (operational unit of the Ministry of Health in charge of health sector policy development for HIV/AIDS)
* National Aids Authority: in charge to lead, manage, coordinate and facilitate the comprehensive and multi-sectoral response to HIV and AIDS in Cambodia
* Ministry of Health
* Key influencer in the MSM and/or TG community
* Key influencer in the EW community
* Khana : an umbrella organization belonging to the HIV/AIDS international Alliance.
* High class and hidden MSM
* Discontinued PrEP user

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — see eligibility criteria
Study Population: MSM, TGW, MEW, FEW will be recruited through community-based organisations, or online, or directly on hotspots.
  PrEP users will be recruited through the pilot program "Khmer PrEP" or online or through community-based organisations or directly on hotspots.
  Health workers will be recruited in HIV services targeting key-populations. Decision makers will be recruited in their organizations respectively.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Knowledge about PrEP | 1 hour
  qualitative assessement
Perception of PrEP | 1 hour
  qualitative assessement
Acceptability of PrEP | 1 hour
  qualitative assessement

SECONDARY OUTCOMES:
To better understand the characteristics, needs and expectations of community-based organisations (CBOs), in order to define the optimal conditions for community-based PrEP implementation | 1 hour
  qualitative assessement
To identify tools that could be useful to increase PrEP awareness and acceptability, especially new technologies (apps, websites) | 1 hour
  qualitative assessement

CONTACTS AND LOCATIONS:
Overall Officials: Vonthanak SAPHONN, Principal Investigator — University of Health Sciences (UHS)
Locations (1):
- University of Health Sciences, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No